CLINICAL TRIAL: NCT00520650
Title: Health Evaluation of Abilify Long-term Therapy
Acronym: HEALTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taiwan Otsuka Pharm. Co., Ltd (Industry)
Responsible Party: Edward C.Y. Peng, Taiwan Otsuka Pharm. Co., Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-06-P01
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
This is a post-market surveillance, and the treatment to patients will be depended upon the decision based on physician's clinical judgment. The health profiles during the switching period, after 12 weeks short-term use, and after 52 weeks long-term use of aripiprazole will be recorded and evaluated.

DETAILED DESCRIPTION:
Further study details as provided by Taiwan Otsuka Pharmaceutical Co., Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the ages of 18 to 65.
2. Having a DSM-IV diagnosis of schizophrenia or schizoaffective disorder.
3. Who are currently taking antipsychotic drugs and clinically intolerable or inadequately controlled that is based upon the clinical judgment of the investigator.

Exclusion Criteria:

1. Pregnant or breast feeding women or planning a pregnancy.
2. Patient received electroconvulsive therapy within 4 weeks before the Screening Visit.
3. A known allergy reaction to any antipsychotic medication (including but not limited to haloperidol, chlorpromazine, thioridazine, pimozide, risperidone, quetiapine, ziprasidone).
4. Patient has clinically relevant organic, neurological, or cardiovascular diseases.
5. Patient has a history of drug or alcohol abuse within the last 12 weeks.
6. Acute psychosis, acute suicidal ideation, or any acute psychiatric condition that might require emergent intervention.
7. Any clinical condition or significant concurrent disease judged by the investigator to complicate the evaluation of the study treatment.
8. Having participated other investigational drug study and taken the investigation drug within one month prior to study entry.
9. Depot neuroleptics should be discontinued at least 2 months prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinical Global Impression-Severity (CGI-S) scale after 52 weeks treatment. | Throughout the study

SECONDARY OUTCOMES:
Change from baseline in CGI-S scale at each visit during the first 39 weeks treatment. | Throughout the study
Change from baseline in total score on the Brief Psychiatric Rating Scale (BPRS) at each visit during the treatment period. | Throughout the study.
Change from baseline in total score on WHOQOL-BREF questionnaire at each visit during the treatment period. | Throughout the study.
Change from baseline in total score on PANSS (optional) questionnaire at each visit during the treatment period. | throughout the study
Change from baseline in total score on SFS (optional) questionnaire at 12 and 52 weeks treatment. | Throughout the study.
Change from Visit 2 on POM questionnaire at each visit during the 12-week switching period. | Throughout the study.
CGI-I scores after 12, 26, 39, and 52 weeks of treatment. | Throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Wen Lin, MD, Principal Investigator — Tri-Service General Hospital
Locations (9):
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital Yun-Lin Branch, Douliu
  - Cardinal Tien Hospital Hsin Chu Mercy Branch, Hsinchu
  - Buddhist Tzu Chi General Hospital, Hualien City
  - Wei Gong Memorial Hospital, Miaoli
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - Tri-Service General Hospital, Taipei